CLINICAL TRIAL: NCT06368817
Title: A Phase II Trial Evaluating Chemotherapy Followed by Response-Based Reduced Radiation Therapy for Patients With Central Nervous System Germinomas
Brief Title: A Study of Lower Radiotherapy Dose to Treat Children With CNS Germinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACNS2321; NCI-2024-03518 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS2321 (Other: Children's Oncology Group); ACNS2321 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2024-04-08; First posted 2024-04-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-02

CONDITIONS: Basal Ganglia Germinoma; Central Nervous System Germinoma; Diabetes Insipidus; Pineal Region Germinoma; Suprasellar Germinoma; Thalamic Germinoma
MeSH Terms: conditions — Germinoma; Diabetes Insipidus | interventions — Radiotherapy, Conformal; Specimen Handling; Carboplatin; Etoposide; Radiotherapy, Intensity-Modulated; Spinal Puncture; Magnetic Resonance Spectroscopy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Stratum I (carboplatin, etoposide, 3D-CRT, IMRT, surgery) (Experimental): See Detailed Description.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Surgical Procedure
- Stratum II (carboplatin, etoposide, 3D-CRT, IMRT) (Experimental): Patients receive carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with localized germinoma achieving PR with normalization of markers who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients undergo MRI and optional blood and tissue sample collection throughout the study. Patients may undergo LP for CSF sample collection during screening and follow up.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Stratum III (carboplatin, etoposide, 3D-CRT, IMRT) (Experimental): Patients receive carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with localized germinoma with normalization of markers who fail to achieve CR or PR who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 24 days. Patients undergo MRI and optional blood and tissue sample collection throughout the study. Patients may undergo LP for CSF sample collection during screening and follow up.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Stratum IV (carboplatin, etoposide, 3D-CRT, IMRT, surgery) (Experimental): Patients receive carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with metastatic germinoma achieving CR undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients with metastatic germinoma and normalization of markers who fail to achieve CR may undergo second-look surgery. Patients found to have mature teratoma or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients undergo MRI and optional blood and tissue sample collection throughout the study. Patients may undergo LP for CSF sample collection during screening and follow up.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Surgical Procedure
- Stratum V (carboplatin, etoposide, 3D-CRT, IMRT) (Experimental): Patients receive carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with metastatic germinoma with normalization of markers who fail to achieve CR who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 24 days. Patients undergo MRI and optional blood and tissue sample collection throughout the study. Patients may undergo LP for CSF sample collection during screening and follow up.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration
- Stratum VI (carboplatin, etoposide, 3D-CRT, IMRT, surgery) (Experimental): Patients receive carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with basal ganglia and thalamic germinoma achieving CR undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients with basal ganglia and thalamic germinoma and normalization of markers who fail to achieve CR may undergo second-look surgery. Patients found to have mature teratoma or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients undergo MRI and optional blood and tissue sample collection throughout the study. Patients may undergo LP for CSF sample collection during screening and follow up.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration; Procedure: Surgical Procedure
- Stratum VII (carboplatin, etoposide, 3D-CRT, IMRT) (Experimental): Patients receive carboplatin IV over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with basal ganglia and thalamic germinoma with normalization of markers who fail to achieve CR who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 24 days. Patients undergo MRI and optional blood and tissue sample collection throughout the study. Patients may undergo LP for CSF sample collection during screening and follow up.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Etoposide; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Lumbar Puncture; Procedure: Magnetic Resonance Imaging; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP 16213; VP-16; VP-16-213; VP-16213; VP16; VP16213
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Lumbar Puncture — Undergo LP
  Other Names: LP; Spinal Tap
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Questionnaire Administration — Ancillary studies
Procedure: Surgical Procedure — Undergo second-look surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery
  Arms: Stratum I (carboplatin, etoposide, 3D-CRT, IMRT, surgery); Stratum IV (carboplatin, etoposide, 3D-CRT, IMRT, surgery); Stratum VI (carboplatin, etoposide, 3D-CRT, IMRT, surgery)

SUMMARY:
This phase II trial studies how well lower dose radiotherapy after chemotherapy (Carboplatin & Etoposide) works in treating children with central nervous system (CNS) germinomas. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Etoposide is in a class of medications known as podophyllotoxin derivatives. It blocks a certain enzyme needed for cell division and DNA repair and may kill cancer cells. Researchers want to see if lowering the dose of standard radiotherapy (RT) after chemotherapy can help get rid of CNS germinomas with fewer long-term side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether 12 Gy whole ventricular irradiation (WVI) and 12 Gy tumor boost would maintain similar efficacy compared to ACNS1123 stratum 2 as measured by event-free survival (EFS) in eligible patients with localized primary central nervous system (CNS) germinoma who present with serum and/or cerebrospinal fluid (CSF) human chorionic gonadotropin-beta (hCGbeta) ≤ 100 IU/L and normal alpha-fetoprotein (AFP), and meet complete response (CR) or continued complete response (CCR) criteria following chemotherapy/second-look surgery (Stratum 1).

SECONDARY OBJECTIVES:

I. To estimate the EFS distribution for patients with localized midline - including bifocal - CNS germinoma with partial response (PR) after chemotherapy, followed by 18 Gy WVI and 12 Gy tumor boost (Stratum 2).

II. To estimate the EFS distribution for patients with localized midline - including bifocal - CNS germinoma with less than a PR after chemotherapy, followed by 24 Gy WVI and 12 Gy tumor boost (Stratum 3).

III. To estimate the overall survival (OS), response rates to chemotherapy and radiotherapy (RT), as well as the patterns of failure of the various cohorts based on tumor characteristics, treatment regimen, and treatment modality.

IV. To determine the impact of tumor characteristics, treatment regimen and treatment modalities on the long-term neuroendocrine function for patients with CNS germinomas.

V. To prospectively evaluate processing speed of children and young adults with CNS germinoma through the Children's Oncology Group (COG) Standardized assessment battery.

EXPLORATORY OBJECTIVES:

I. To estimate the EFS distribution for patients with metastatic germinomas treated with chemotherapy followed by craniospinal irradiation (CSI) [18 Gy for CR/CCR (Stratum 4)] or [24 Gy for less than CR (Stratum 5)] with a 12 Gy tumor boost to the pre-treatment volume, including metastatic sites.

II. To estimate the EFS distribution for patients with basal ganglia and thalamic germinomas (BGTG) treated with chemotherapy followed by whole brain irradiation (WBI) [18 Gy for CR/CCR (Stratum 6)] or [24 Gy for less than CR (Stratum 7)] with a 12 Gy tumor boost to the pre-treatment volume.

III. To prospectively collect blood, cerebrospinal fluid, and tumor tissue at diagnosis and second-look surgery (if feasible) for future biology studies.

IV. To prospectively measure the incidence of cerebral vascular events (stroke or transient ischemic attacks) in the follow-up period and longitudinally evaluate and model the cognitive, social and behavioral functioning of children and young adults with CNS germinoma through the COG Standardized assessment battery, and compare these outcomes based on tumor characteristics, treatment regimen, and treatment modality.

OUTLINE:

INDUCTION PHASE: All patients receive carboplatin intravenously (IV) over 15-60 minutes on day 1 and etoposide IV over 90-120 minutes on days 1-3 of each cycle. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity.

Patients are then assigned to 1 of 7 strata.

STRATUM I: Patients with localized germinoma achieving CR with normalization of markers undergo 3-dimensional conformal radiation therapy (3DCRT) or intensity-modulated radiation therapy (IMRT) once daily (QD) 5 days a week for 16 days. Patients achieving PR with normalization of markers may undergo second-look surgery. Patients found to have mature teratoma or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 16 days. Patients with normalization of markers who fail to achieve CR or PR may undergo second-look surgery. Patients found to have mature teratoma or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 16 days. Patients with bifocal germinoma undergo 3DRT or IMRT QD 5 days a week for 16 days.

STRATUM II: Patients with localized germinoma achieving PR with normalization of markers who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 20 days.

STRATUM III: Patients with localized germinoma with normalization of markers who fail to achieve CR or PR who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 24 days.

STRATUM IV: Patients with metastatic germinoma achieving CR undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients with metastatic germinoma and normalization of markers who fail to achieve CR may undergo second-look surgery. Patients found to have mature teratoma or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 20 days.

STRATUM V: Patients with metastatic germinoma with normalization of markers who fail to achieve CR who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 24 days.

STRATUM VI: Patients with basal ganglia and thalamic germinoma achieving CR undergo 3DRT or IMRT QD 5 days a week for 20 days. Patients with basal ganglia and thalamic germinoma and normalization of markers who fail to achieve CR may undergo second-look surgery. Patients found to have mature teratoma or non-viable tumor undergo 3DRT or IMRT QD 5 days a week for 20 days.

STRATUM VII: Patients with basal ganglia and thalamic germinoma with normalization of markers who fail to achieve CR who do not undergo second-look surgery undergo 3DRT or IMRT QD 5 days a week for 24 days.

Patients with non-normalized tumor markers or PD and no second-look surgery or viable tumor during second-look surgery discontinue protocol therapy.

All patients undergo magnetic resonance imaging (MRI) and optional blood and tissue sample collection throughout the study. Patients may undergo lumbar puncture (LP) for CSF sample collection during screening and follow up.

After completion of study treatment, patients are followed up every 3 months for 12 months, every 4 months for 24 months, and then annually for up to 120 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 3 years and < 30 years at the time of study enrollment
* Patients must be newly-diagnosed primary localized germinoma of the suprasellar and/or pineal region by pathology and/or serum and/or CSF hCGbeta 5-50 mIU/mL AND institutional normal AFP (or ≤ 10 ng/mL if no institutional normal exists), including tumors with contiguous ventricular or unifocal parenchymal extension. No histologic confirmation required
* Patients with EITHER (A) bifocal (pineal + suprasellar) involvement OR (B) pineal lesion with diabetes insipidus (DI) AND hCGbeta ≤ 100 mIU/mL in serum and/or CSF AND institutional normal AFP (or ≤ 10 ng/mL if no institutional normal exists) in both serum and CSF. No histologic confirmation required
* Patients with hCGbeta 51-100 mIU/mL in serum and/or CSF and institutional normal AFP (or ≤ 10 ng/mL if no institutional normal exists) in both serum and CSF. Histologic confirmation of germinoma IS required
* Patients with germinoma of the basal ganglia and or/thalamic primary sites are eligible
* Patients with metastatic germinoma including non-contiguous disease or distant disease in the brain, ventricles, or spine are eligible
* Patients with germinoma admixed with mature teratoma are eligible
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age
* Patients must have eligibility confirmed by Rapid Central Imaging Review performed on APEC14B1-CNS
* Imaging studies must be obtained within 31 days prior to study enrollment and start of protocol therapy. (Note: for patients that have had surgery and post-operative imaging performed, it is the post-operative MRI that must be obtained within 31 days prior to enrollment.)
* Patients must have a cranial magnetic resonance imaging (MRI) with and without gadolinium at diagnosis/prior to enrollment. If surgical resection is performed, patients must have pre-operative and post-operative brain MRI with and without gadolinium. The post-operative brain MRI should be obtained within 72 hours of surgery. If patient has a biopsy only, post-operative brain MRI is recommended but not required
* Patients must have a spine MRI with gadolinium obtained at diagnosis/prior to enrollment
* Patients must be enrolled, and protocol therapy must begin, no later than 31 days after definitive surgery or clinical diagnosis, whichever is later
* Patients must have eligibility confirmed by Rapid Central Tumor Marker Review performed on APEC14B1-CNS
* Lumbar CSF must be obtained prior to study enrollment unless medically contraindicated. If a patient undergoes surgery and lumbar CSF cytology cannot be obtained at the time of surgery, then it should be performed at least 10 days following surgery and prior to study enrollment. False positive cytology can occur within 10 days of surgery. Of note, lumbar CSF should not be performed prior to obtaining spine MRI, as this can make interpretation of the spine MRI less clear
* Patients must have CSF tumor markers obtained prior to study enrollment unless medically contraindicated. Ventricular CSF obtained at the time of CSF diversion procedure (if performed) is acceptable for tumor markers but lumbar CSF is preferred. In case CSF diversion and biopsy/surgery are combined, CSF tumor markers should be collected first. Ideally serum and CSF tumor markers should be collected at the same time and processed without delay
* For patients with solid tumors: Peripheral absolute neutrophil count (ANC) >= 1000/uL (Must be performed within 7 days prior to enrollment unless otherwise indicated)
* For patients with solid tumors: Platelet count >= 100,000/uL (transfusion independent) (Must be performed within 7 days prior to enrollment unless otherwise indicated)
* For patients with solid tumors: Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) (Must be performed within 7 days prior to enrollment unless otherwise indicated)
* For pediatric patients (age 3-17 years): A serum creatinine based on age/gender as follows (Must be performed within 7 days prior to enrollment unless otherwise indicated):

  * Age: 3 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male); 0.8 (female)
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): 1 (male); 1 (female)
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: ≥ 17 years; maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female) OR a 24-hour urine creatinine clearance ≥ 70 mL/min/1.73 m^2 OR a glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard).
  * Note: Estimated GFR (eGFR) from serum or plasma creatinine, cystatin C or other estimates are not acceptable for determining eligibility.
  * For adult patients (age 18 years or older) (Must be performed within 7 days prior to enrollment unless otherwise indicated):

    * Creatinine clearance ≥ 70 mL/min, as estimated by the Cockcroft and Gault formula or a 24-hour urine collection. The creatinine value used in the calculation must have been obtained within 28 days prior to registration. Estimated creatinine clearance is based on actual body weight
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age (Must be performed within 7 days prior to enrollment unless otherwise indicated)
* Serum glutamic-pyruvic transaminase (SGPT) (alanine transaminase [ALT]) ≤ 135 U/L (Must be performed within 7 days prior to enrollment unless otherwise indicated)

  * Note: For the purpose of this study, the ULN for SGPT (ALT) has been set to the value of 45 U/L
* No evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% if there is clinical indication for determination
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* CNS toxicity =< grade 2
* Patients must not be in status epilepticus, coma or assisted ventilation prior to study enrollment
* HIV-infected patients on effective anti-retroviral therapy with undetectable viral load are eligible for this study

Exclusion Criteria:

* Patients with any of the following malignant pathological elements are not eligible:

  * Endodermal sinus (yolk sac)
  * Embryonal carcinoma, choriocarcinoma
  * Malignant/immature teratoma and mixed germ cell tumor (GCT) (i.e., may include some germinoma)
* Patients with only mature teratoma upon tumor sampling at diagnosis and negative tumor markers are not eligible
* Patients who have received any prior tumor-directed therapy for their diagnosis of germinoma other than surgical intervention and corticosteroids are not eligible
* Female patients who are pregnant since fetal toxicities and teratogenic effects have been noted for several of the study drugs. A pregnancy test is required for female patients of childbearing potential.

  * Note: Serum and urine pregnancy tests may be falsely positive due to HCGbeta-secreting germ cell tumors. Ensure the patient is not pregnant by institutional standards
* Lactating females who plan to breastfeed their infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Ages: 3 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2033-11-04 (Estimated); Study Completion 2033-11-04 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) (Stratum I) | Evaluated at 2- and 3-years post-radiation initiation
  Will be estimated for eligible and evaluable patients assigned to Stratum 1 using Kaplan-Meier (KM) EFS estimates at 2 and 3 years with respective 80% two-sided confidence intervals. Time from initiation of radiation to the first occurrence of any of the following events: biochemical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause.

SECONDARY OUTCOMES:
EFS (Stratum II) | Evaluated at 2- and 3-years post-radiation initiation
  Will be estimated for eligible and evaluable patients assigned to Stratum 2 using KM methods at 2 and 3 years with respective 80% two-sided confidence intervals. Time from initiation of radiation to the first occurrence of any of the following events: biochemical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause.
EFS (Stratum III) | Evaluated at 2- and 3-years post-radiation initiation
  Will be estimated for eligible and evaluable patients assigned to Stratum 3 using KM methods at 2 and 3 years with respective 80% two-sided confidence intervals. Time from initiation of radiation to the first occurrence of any of the following events: biochemical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause.
Radiographic response rate | Following the completion of Induction therapy, approximately 12 weeks post-chemotherapy initiation
  Will report the response rates using the respective sample proportions and exact binomial two-sided 95% confidence intervals.
Marker tumor response rate | Following the completion of Induction therapy, approximately 12 weeks post-chemotherapy initiation
  Will report the response rates using the respective sample proportions and exact binomial two-sided 95% confidence intervals.
Overall survival (OS) | Time from initiation of radiation therapy until death by any cause, up to 10 years post-enrollment
  Will use KM methods to estimate stratum-specific OS.
Neuroendocrine dysfunction (including growth hormone deficiency) | Time from initiation of RT until date of diagnosis of neuroendocrine dysfunction event, up to 10 years post-enrollment
  Will be summarized by the Kalbfleisch-Prentice cumulative incidence function (CIF) approach, separately by stratum and by neuroendocrine dysfunction event. Competing risks will include disease progression and death, and patients without events or competing risks will be censored at the time of their last follow-up.
Processing speed | At 9 months (+/- 3 months), 30 months (+/- 3 months), and 60 months (+/- 3 months) after diagnosis
  Will be assessed by processing speed index tasks for the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (WPPSI-IV), Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V) or Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) depending on age. The mean processing speed at 30-months post-diagnosis in ACNS2321 Stratum 1 patients will be compared to the respective mean in ACNS1123 Stratum 2 patients who had a CR/CCR and received 18 Gy WVI + 12 Gy boost to primary site.

OTHER OUTCOMES:
EFS (Stratum IV and Stratum V) | Evaluated at 2- and 3-years post-radiation initiation
  Will be estimated separately for eligible and evaluable patients assigned to Stratum 4 and 5 using KM methods at 2 and 3 years with respective 80% two-sided confidence intervals. Time from initiation of radiation to the first occurrence of any of the following events: biochemical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause.
EFS (Stratum VI and Stratum VII) | Evaluated at 2- and 3-years post-radiation initiation
  Will be estimated separately for eligible and evaluable patients assigned to Stratum 6 and 7 using KM methods at 2 and 3 years with respective 80% two-sided confidence intervals. Time from initiation of radiation to the first occurrence of any of the following events: biochemical or radiographic disease progression, disease recurrence, second malignant neoplasm, or death from any cause.
Incidence of cerebral vascular events (stroke or transient ischemic attacks) | Up to 10 years post-enrollment
  Will be reported as the number of cerebral vascular events.
Working memory | At 9 months (+/- 3 months), 30 months (+/- 3 months), and 60 months (+/- 3 months) after diagnosis
  Will be assessed by Wechsler Intelligence Scale for Children - Fifth Edition (WISC-V) or Wechsler Adult Intelligence Scale - Fourth Edition (WAIS-IV) Digit Span subtest depending on age. Mean scores over time will be computed for each stratum.
Verbal learning | At 9 months (+/- 3 months), 30 months (+/- 3 months), and 60 months (+/- 3 months) after diagnosis
  Will be assessed by California Verbal Learning Test - Children's Version for 5 years through 17 years or California Verbal Learning Test - Third for ages 17 and up depending on age. Mean scores over time will be computed for each stratum.
Patient-reported outcome measures of executive function | At 9 months (+/- 3 months), 30 months (+/- 3 months), and 60 months (+/- 3 months) after diagnosis
  Will be assessed by the Behavioral Rating Inventory of Executive Function (BRIEF-2 and BRIEF-A) depending on patient's age. Mean scores over time will be computed for each stratum.
Health-reported quality of life | At 9 months (+/- 3 months), 30 months (+/- 3 months), and 60 months (+/- 3 months) after diagnosis
  Will be assessed by the PedsQL 4.0 Generic Module. Mean scores over time will be computed for each stratum.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Abdelbaki, Principal Investigator — Children's Oncology Group
Locations (102):
- United States (87):
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Albany Medical Center, Albany, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Australia (5):
  - John Hunter Children's Hospital, Hunter Regional Mail Centre, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - CHU de Quebec-Centre Hospitalier de l'Universite Laval (CHUL), Québec